CLINICAL TRIAL: NCT01179126
Title: Complete Revascularization Or streSS Echo in Patients With Multivessel Disease and ST-segment Elevation Acute Myocardial Infarction
Brief Title: Strategies of Revascularization in Patients With ST-segment Elevation Myocardial Infarction (STEMI) and Multivessel Disease
Acronym: CROSS-AMI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Complexo Hospitalario Universitario de A Coruña (Other)
Responsible Party: Principal Investigator, Rodrigo Estévez-Loureiro, MD, PhD, Complexo Hospitalario Universitario de A Coruña
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CROSS-AMI
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Myocardial Infarction; Angioplasty, Transluminal, Percutaneous Coronary; Echocardiography, Stress
Keywords: myocardial infarction; primary angioplasty; multivessel disease; stress echocardiography
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- complete multivessel revascularization (Experimental)
  Interventions: Procedure: complete multivessel revascularization
- stress echo guided revascularization (Active Comparator)
  Interventions: Procedure: stress echocardiography and revascularization if required

INTERVENTIONS:
Procedure: complete multivessel revascularization — After a successful primary PCI these patients will undergo complete revascularization of non-culprit lesions in a staged procedure during the index admission
  Arms: complete multivessel revascularization
Procedure: stress echocardiography and revascularization if required — after successful primary PCI, this group will undergo a stress echo to evaluate the significance of non-culprit lesions. If large area of ischemia is demonstrated, the artery supplying that are will be revascularized.
  Arms: stress echo guided revascularization

SUMMARY:
Multivessel disease has been reported to occur between 40 and 60% of patients with ST-segment elevation myocardial infarction (STEMI) and has been associated to a worse prognosis. Multivessel revascularization offers a myriad of potential advantages as enhance of the collateral blood flow, greater myocardial salvage, the stabilization of other lesions that can be potentially vulnerable, and the achievement of a complete revascularization, factor that is associated with a better prognosis. On the other hand, the prolongation of procedural duration, the hazard of contrast induced nephropathy and the peri-procedural complications can limit the widespread of this practice.

To date, very few observational studies have focused in the multivessel revascularization with disparity of results. Whereas ones have observed an increase of adverse cardiovascular events and thus not recommend it, others have shown neutral results.

Stress echocardiography has been shown to be an adequate technique for the diagnosis of coronary artery disease and could be an appropriate tool for selecting the lesions that need to be revascularized because they induce large areas of ischemia. However, this technique has also limitations like the high operator-dependence.

Therefore, the investigators sought to study if the complete multivessel revascularization of patients with STEMI treated by means of primary percutaneous coronary intervention (PCI) has an impact on prognosis compared to a strategy of treating only those non-culprit lesions that produce large areas of ischemia in a stress test.

ELIGIBILITY:
Inclusion Criteria:

* Typical chest pain lasting >30 minutes with ST-segment elevation >=1mm in >=2 contiguous ECG leads or left bundle branch block and presentation < 48 hours since symptom onset.
* Patients undergoing rescue PCI
* Patients with effective lysis and coronary angiography in less than 24 hours
* Presence of other lesion >=70% in a non-culprit artery.
* Informed consent

Exclusion Criteria:

* Significant left main disease
* Lesions in vessels < 2 mm
* Lesions in branches of a main epicardial coronary artery and short irrigation territory
* Previous coronary artery bypass graft (CABG)
* Any coronary intervention in the previous month
* Cardiogenic shock
* Anatomic features no suitable for coronary intervention
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-09; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Combined event of cardiovascular death/re-myocardial infarction/revascularization of any vessel/admission due to heart failure | one year

SECONDARY OUTCOMES:
Incidence of acute renal failure (contrast induced nephropathy) | Admission
Cost analysis of both strategies | 1 year
Death | one year
  cardiovascular death
re-myocardial infarction | one year
revascularization of any vessel | one year
admission due to heart failure | one year

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Estevez-Loureiro, MD, Principal Investigator — Interventional Cardiology. Complejo Hospitalario Universitario A Couna; Ramon Calvino-Santos, MD, Study Chair — Interventional Cardiology. Complejo Hospitalario A Couna; Nicolas Vazquez-Gonzalez, MD, Study Chair — Interventional Cardiology. Complejo Hospitalario A Couna; Jorge Salgado-Fernandez, MD, Study Chair — Interventional Cardiology. Complejo Hospitalario A Couna; Pablo Pinon-Esteban, MD, Study Chair — Interventional Cardiology. Complejo Hospitalario A Couna; Guillermo Aldama-Lopez, MD, Study Chair — Interventional Cardiology. Complejo Hospitalario A Couna; Xacobe Flores-Rios, MD, Study Chair — Interventional Cardiology. Complejo Hospitalario A Couna; Jesus Peteiro, MD, PhD, Study Chair — Stress Echo Unit. Complejo Hospitalario A Couna; Alberto Bouzas-Mosquera, MD, Study Chair — Stress Echo Unit. Complejo Hospitalario A Couna; Jose Angel Rodriguez-Fernandez, MD, Study Chair — Coronary Care Unit. Complejo Hospitalario A Couna
Locations (1):
- Complejo Hospitalario Universitario A Coruna, A Coruña, A Coruna, Spain

REFERENCES:
- [Derived] Flores-Rios X, Calvino-Santos RA, Estevez-Loureiro R, Peteiro-Vazquez J, Salgado-Fernandez J, Rodriguez-Vilela A, Franco-Gutierrez R, Bouzas-Mosquera A, Rodriguez-Fernandez JA, Marzoa-Rivas R, Gonzalez-Juanatey C, Aldama-Lopez G, Pinon-Esteban P, Vazquez-Gonzalez N, Muniz-Garcia J, Vazquez-Rodriguez JM. Economic evaluation of complete revascularization versus stress echocardiography-guided revascularization in the STEACS with multivessel disease. Rev Esp Cardiol (Engl Ed). 2021 Dec;74(12):1054-1061. doi: 10.1016/j.rec.2020.09.028. Epub 2020 Nov 27. English, Spanish. PMID 33257214
- [Derived] Calvino-Santos R, Estevez-Loureiro R, Peteiro-Vazquez J, Salgado-Fernandez J, Rodriguez-Vilela A, Franco-Gutierrez R, Bouzas-Mosquera A, Rodriguez-Fernandez JA, Mesias-Prego A, Gonzalez-Juanatey C, Aldama-Lopez G, Pinon-Esteban P, Flores-Rios X, Soler-Martin R, Seoane-Pillado T, Vazquez-Gonzalez N, Muniz J, Vazquez-Rodriguez JM. Angiographically Guided Complete Revascularization Versus Selective Stress Echocardiography-Guided Revascularization in Patients With ST-Segment-Elevation Myocardial Infarction and Multivessel Disease: The CROSS-AMI Randomized Clinical Trial. Circ Cardiovasc Interv. 2019 Oct;12(10):e007924. doi: 10.1161/CIRCINTERVENTIONS.119.007924. Epub 2019 Sep 26. PMID 31554422